CLINICAL TRIAL: NCT01893723
Title: Analgesia Nociception Index Guided Remifentanil Administration During Propofol Anesthesia for Laparoscopic Surgery : Multicenter Randomized Clinical Trial
Brief Title: Analgesia Nociception Index Guided Remifentanil Administration During Propofol Anesthesia for Laparoscopic Surgery
Acronym: AIVOC-ANI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes of usual clinical practices
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2010_51; 2011-A00947-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2013-06-18; First posted 2013-07-09 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: General Anesthesia
Keywords: autonomous nervous system monitoring; analgesia nociception balance; remifentanil; analgesia nociception index; hemodynamic reactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ANI guided remifentanil arm (Experimental): remifentanil targets are increased or decreased depending on ANI readings. In case of high blood pressure associated with elevated ANI, nicardipine is administered.
  Interventions: Procedure: ANI guided remifentanil
- ANI blind arm (Other): remifentanil target is adapted as is usual during general anesthesia, depending on hemodynamic reactions to nociceptive surgical stimulations. In case of elevated blood pressure despite a maximum target of 10 ng/ml (Minto Pk/pD model), then nicardipine is administered.
  Interventions: Procedure: ANI blind arm

INTERVENTIONS:
Procedure: ANI guided remifentanil — remifentanil administration during propofol anesthesia for laparoscopic surgery is ANI guided
  Arms: ANI guided remifentanil arm
Procedure: ANI blind arm — remifentanil administration during propofol anesthesia for laparoscopic surgery is not ANI guided
  Arms: ANI blind arm

SUMMARY:
The Physiodoloris (MetroDoloris, Lille, France) monitor, CE marqued, uses the ECG signal in order to compute the Analgesia Nociception Index (ANI) which has been shown to measure the relative parasympathetic tone, and hence to reflect the analgesia/nociception balance during general anesthesia. The primary endpoint of this randomized multicenter study is to measure whether there is a benefit to use the ANI in order to adapt remifentanil administration during propofol anesthesia for laparoscopic surgery. Primary endpoint : lesser proportion of patients presenting with at least one episode of hemodynamic reactivity, hypotension or bradycardia in the ANI guided group vs control group ?

DETAILED DESCRIPTION:
The Physiodoloris (MetroDoloris, Lille, France) monitor, CE marqued, uses the ECG signal in order to compute the Analgesia Nociception Index (ANI) which has been shown to measure the relative parasympathetic tone, and hence to reflect the analgesia/nociception balance during general anesthesia. The primary endpoint of this randomized multicenter study is to measure whether there is a benefit to use the ANI in order to adapt remifentanil administration during propofol anesthesia for laparoscopic surgery. Primary endpoint is: lesser proportion of patients presenting with at least one episode of hemodynamic reactivity, hypotension or bradycardia in the ANI guided group vs control group ?

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic cholecystectomy or gynecological laparoscopic surgery
* ASA I or II
* adult patient
* body mass index between 17 and 33 kg/m2

Exclusion Criteria:

* pregnancy
* arrhythmia
* pace maker
* diabetes mellitus
* dysautonomia
* treatment with beta blocking agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients presenting at least once with hemodynamic reactivity, hypotension or bradycardia | end of surgery (around 60 to 90 min after start)

SECONDARY OUTCOMES:
total administered remifentanil | end of surgery
number of target changes | end of surgery (around 60 to 90 min after start)
morphine sulfate total administration after end of surgery | during two hours after end of surgery
Visual Analog Scale evaluation of pain after surgery | during two hours after end of surgery
ANI measure during surgery | from start to end of surgery (around 60 to 90 min)
number of bradycardia and hypotension | from start to end of surgery (around 60 to 90 min )
total administered dose of ephedrine | between start and end of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu JEANNE, MD, Principal Investigator — University Hospital, Lille
Locations (5):
- University Hospital Erasme (ULB), Brussels, Belgium
- France (4):
  - Clinique privée d'ANTONY, Antony
  - University Hospital Claude Huriez, Lille
  - University Hospital Roger Salengro, Lille
  - University Hospital, Saint-Etienne